CLINICAL TRIAL: NCT00153803
Title: A National Web-Based Randomized Phase III Study of Erlotinib or Placebo Following Concurrent Docetaxel, Carboplatin, and Thoracic Radiotherapy in Patients With Inoperable Stage III Non-Small Cell Lung Cancer (D0410).
Brief Title: Erlotinib or Placebo Following Chemoradiotherapy (Chemo/RT) in Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sanofi (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-0410
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-small Cell Lung Cancer; NSCLC
Keywords: Erlotinib; Tarceva; Web based; Stage III NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Erlotinib (Tarceva) 150mg: Erlotinib 150mg orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events, death or completion of 3 years of therapy.
  Interventions: Drug: Erlotinib (tarceva)
- 2 (Placebo Comparator): Matched Placebo: Matched placebo orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events death or completion of 3 years of therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib (tarceva) — Erlotinib 150mg orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events, death or completion of 3 years of therapy.
  Arms: 1
Drug: Placebo — Matched placebo orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events death or completion of 3 years of therapy.
  Arms: 2

SUMMARY:
This is a national, randomized, web-based, double-blind study to determine whether erlotinib (Tarceva) compared to placebo improves progression-free survival (PFS) for patients with inoperable, stage III NSCLC following concurrent docetaxel, carboplatin and thoracic radiotherapy. We hypothesize that the introduction of this orally active, well-tolerated agent following concurrent chemoradiation and prior to the emergence of drug resistance will prolong the progression-free survival by 40% (10 months → 14 months).

DETAILED DESCRIPTION:
The promising activity of erlotinib as a single agent in advanced refractory NSCLC along with its oral administration and favorable adverse event profile makes this agent an excellent candidate to incorporate into combined modality therapy in the early stages of lung cancer. Based on these data, erlotinib is an attractive novel approach to maintenance therapy in unresectable stage III NSCLC following completion of concomitant chemoradiation. Although, a subset of patients with unresectable stage III NSCLC will be long-term survivors following chemotherapy and thoracic radiation therapy, the vast majority relapse within the first year following therapy and eventually die from chemotherapy refractory disease. We hypothesize that the introduction of an potent tyrosine kinase inhibitor to the epidermal growth factor receptor following effective concomitant chemoradiotherapy with docetaxel and carboplatin will prolong the progression-free survival time for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, stage IIIA or IIIB NSCLC (measurable disease is not required)
* No evidence of metastatic disease
* No prior treatment
* Adequate organ function
* Adequate pulmonary function (FEV >= 1.0L or predicted FEV >0.8L)

Exclusion Criteria:

* Metastasis
* Prior treatment
* Malignant pleural or pericardial effusion
* Peripheral neuropathy >= grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2005-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Study Chair — Norris Cotton Cancer Center
Locations (65):
- United States (65):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Oncology Specialties, P.C., Huntsville, Alabama
  - Cooper Clinic, Fort Smith, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Northstate Cancer Speciality, Redding, California
  - Mercy General Hospital, Sacramento, California
  - St. Francis Hospital Cancer Center, Hartford, Connecticut
  - Connecticut Oncology Group, Middletown, Connecticut
  - George Bray Cancer Center/New Britain General Hospital, New Britain, Connecticut
  - Oncology and Hematology Associates, PC, New London, Connecticut
  - Whittingham Cancer Center at Norwalk Hospital, Norwalk, Connecticut
  - Hematology/Oncology PC/Carl and Dorothy Bennet Cancer Center, Stamford, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Pasco Hernando Oncology Associates, Brooksville, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Lee Cancer Clinic, Fort Myers, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Cancer Care of North Florida, Lake City, Florida
  - Pasco/Hernando Oncology, New Port Richey, Florida
  - Mid Florida Oncology, Orange City, Florida
  - MD Anderson, Orlando, Florida
  - Oncology & Hematology Association of West Broward, Tamarac, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Joliet Hematology Associates, Joliet, Illinois
  - Investigative Clinical Research of Indiana LLC, Indianapolis, Indiana
  - Howard Regional Health System, Kokomo, Indiana
  - McFarland Clinic, Ames, Iowa
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Western Hematology Oncology, Paducah, Kentucky
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Harbor View Cancer Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Frederick Smith, MD, Chevy Chase, Maryland
  - Community Hematology Oncology, Olney, Maryland
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Fallon Clinic Hematology/ Oncology, Worcester, Massachusetts
  - Bay Medical Cancer Center, Bay City, Michigan
  - Southeast Nebraska Hematology/Oncology, Lincoln, Nebraska
  - Methodist Cancer Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth-Hitchcock-Keene, Keene, New Hampshire
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Sussex County Medical Associates, Newton, New Jersey
  - Queens Medical Associates, Fresh Meadows, New York
  - Winthrop University Hospital, Mineola, New York
  - Hematology Oncology Associates of Rockland, PC, New York, New York
  - Lincoln Hospital, The Bronx, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Aultman Cancer Center, Canton, Ohio
  - The Cleveland Clinic Foundation Hematology/Med Oncology, Cleveland, Ohio
  - Legacy Good Samaritan, Portland, Oregon
  - SCOA-SC Onc Assoc, Columbia, South Carolina
  - VA Department of Hematology/Oncology, Houston, Texas
  - Hope Oncology, Richardson, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Tyler Hematology/Oncology, Tyler, Texas
  - Veterans Administration Medical Center, White River Junction, Vermont
  - Virginia Oncology Associates Research Program, Newport News, Virginia
  - Olympic Hematology/Oncology, Bremerton, Washington
  - Morgantown Internal Medicine Group, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1: 245 patients were registered & randomized. Of those, 10 patients were ineligible due to incorrect stage, withdrawal of consent, inability to meet radiation therapy parameters, and inadequate functional status. The number of participants for each specific reason for ineligibility is unknown. They did not receive any study intervention.
Pre-assignment Details: Period 2:Study drug dispensed to only chemoradiation patients who did not experience disease progression, consent withdrawal, death, investigators discretion, or toxicity.
Groups:
- Tarceva: Tarceva 150mg
  Erlotinib (tarceva): Erlotinib 150mg orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events, death or completion of 3 years of therapy.
- Placebo: Matched Placebo
  Placebo: Matched placebo orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events death or completion of 3 years of therapy.
Period: Concurrent Chemoradiation
Arm/Group | Tarceva | Placebo
Started (Patients randomized) | 123 | 122
Received Chemoradiation | 118 | 117
Completed | 118 | 117
Not Completed | 5 | 5
Period: Investigational Drug
Arm/Group | Tarceva | Placebo
Started (Patients who participated in Period 1) | 118 | 117
Investigational Drug Dispensed | 77 | 75
Completed (Received at least one dose) | 77 | 75
Not Completed | 41 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tarceva | Placebo | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Continuous [Median (Full Range); unit: years] | 68 [39 to 89] | 67 [38 to 84] | 67.5 [38 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 55 | 100
  Male | 78 | 67 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 109 | 106 | 215
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as time from randomization until documented disease progression or death from any cause. The Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.0) was used to determine disease progression. Irradiated target lesions were considered non-measurable disease. Symptomatic radiographic changes of irradiated non-measurable disease required pathologically confirmation or positive FDG-PET scan 6 months following completion of concurrent chemoradiation to be considered locoregional disease progression. Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression was considered distant disease progression.
Time Frame: 5 years
Population: NA = not available; The data cannot be located/provided due to the PI leaving the institution.
Measure: Median (Full Range); unit: Months
Arm/Group | Tarceva | Placebo
Number analyzed (Participants) | 118 | 117
Months | 7.4 [NA to NA] — Data could not be found; The data cannot be located/provided due to the PI leaving the institution. | 8.1 [NA to NA] — Data could not be found; The data cannot be located/provided due to the PI leaving the institution.
Statistical Analysis 1: Comparison: Tarceva vs Placebo; Test type: Superiority; p = 0.165, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.65 to 1.33]

2. Secondary Outcome: Overall Survival
Time Frame: From date of randomization until the date of death from any cause, assessed up to 50 months
Population: NA = not available; The data cannot be located/provided due to the PI leaving the institution.
Measure: Median (Full Range); unit: Months
Groups:
- Tarceva: Tarceva 150mg
  Erlotinib (tarceva): Erlotinib 150mg orally each day. Patients will be treated on a continuous, once daily oral dosing schedule until disease progression, withdrawal of consent, unacceptable adverse events, death or completion of 2 years of therapy.
Arm/Group | Tarceva | Placebo
Number analyzed (Participants) | 118 | 117
Months | 16.5 [NA to NA] — Data could not be found; The data cannot be located/provided due to the PI leaving the institution. | 20.3 [NA to NA] — Data could not be found; The data cannot be located/provided due to the PI leaving the institution.
Statistical Analysis 1: Comparison: Tarceva vs Placebo; Test type: Superiority; p = 0.32, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.85 to 1.63]

3. Secondary Outcome: Percent of Participants Surviving 3 Years
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Tarceva | Placebo
Number analyzed (Participants) | 118 | 117
percentage of participants | 37 | 41

4. Secondary Outcome: Serious Adverse Event Profile Relating to Death, Disability, Life-threatening, Hospitalization, and Impairment/Damage for Concurrent Chemoradiation
Description: Number of participants with treatment-related serious adverse events (SAEs) observed in each SAE category for each arm relating to death, disability, life-threatening, hospitalization, and impairment/damage is reported. For participants with multiple SAEs, the SAE report having the strongest relationship to study drug is summarized.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tarceva | Placebo
Number analyzed (Participants) | 118 | 117
Participants
  Death | 7 | 6
  Disability | 0 | 0
  Life-threatening | 2 | 4
  Hospitalization | 26 | 36
  Impairment/damange | 3 | 3
  Other | 1 | 0

5. Secondary Outcome: Serious Adverse Event Profile Relating to Death, Disability, Life-threatening, Hospitalization, and Impairment/Damage for Erlotinib and Placebo
Description: as for outcome 4
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tarceva | Placebo
Number analyzed (Participants) | 77 | 75
Participants
  Death | 10 | 6
  Disability | 0 | 0
  Life-threatening | 1 | 1
  Hospitalization (initial or prolonged) | 30 | 23
  Impairment/damange | 2 | 1
  Other | 1 | 0

ADVERSE EVENTS:
Time Frame: The intent-to-treat population included 235 eligible randomized patients to the erlotinib arm (n = 118) or placebo arm (n = 117); 245 randomized, 10 became ineligible prior to any treatment. Patients were evaluated with a medical history, physical exam, laboratory studies, and toxicity assessment starting at 1st dose, every 4 weeks for 2 months, then every 8-12 weeks until treatment discontinuation. Participants were evaluated, on average, for 6 months, and through study completion up to 3 years
Description: Common Toxicities are reported. Adverse events (Serious, Other Adverse Events) are reporting for only those participants who are included in the intent-to-treat population .This study used the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0 for grading and reporting of toxicities and adverse events.
Arm/Group | Chemoradiation Before Tarceva | Chemoradiation Before Placebo | Tarceva | Placebo
All-Cause Mortality (participants affected / at risk) | 26/118 | 27/117 | 43/77 | 40/75
Serious Adverse Events (participants affected / at risk) | 36/118 | 38/117 | 39/77 | 23/75
Other Adverse Events (participants affected / at risk) | 12/118 | 8/117 | 8/77 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation Before Tarceva (N=118) | Chemoradiation Before Placebo (N=117) | Tarceva (N=77) | Placebo (N=75)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) — Supraventricular and nodal arrhythmia
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac General (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) — Cardiac General
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Cardiac ischemia/infarction
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ventricular arrhythmia
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Fistula, Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Gastritis (including bile reflux gastritis)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis/stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Mucositis/stomatitis (functional/symptomatic) Esophagus
Perforation, GIColon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — GI/Colon Perforation
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constitutional Symptoms - Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Fatigue (asthenia, lethargy, malaise)
Constitutional Symptoms - Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10eFever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)9/L)
Constitutional Symptoms- Other (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage - Respiratory tract NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hemorrhage, pulmonary/upper respiratory/ Respiratory tract None otherwise specified (NOS)
Hemorrhage, GI Lower (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hemorrhage, pulmonary/upper respiratory Bronchopulmonary
Hemorrhage, pulmonary/upper respiratory- Lung (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Hemorrhage, pulmonary/upper respiratory- Lung
Hemorrhage/Bleeding - Other (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Abdomen NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — None otherwise specified (NOW)
Pain - Bone (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain - Joint (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain- Chest/thorax (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Allergic reaction/hypersensitivity (including drug fever)
Colitis, Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — example: Clostridium difficile
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection - Blood (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Infection with normal ANC or Grade 1 or 2 neutrophils Blood
Infection - Foreign body (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Infection with normal ANC or Grade 1 or 2 neutrophils Foreign body (e.g., graft, implant, prosthesis, stent)
Infection - Lung (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) — Infection with normal ANC or Grade 1 or 2 neutrophils Lung (pneumonia)
Infection - Other (Infections and infestations) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Infection - Wound (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Infection with normal ANC or Grade 1 or 2 neutrophils Wound
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal / Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Musculoskeletal / Soft Tissue - Other
Cerebrovascular Ischemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurology - Other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction - Ureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) | 4 (4)
Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-operative Injury - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Vascular - Other (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation Before Tarceva (N=118) | Chemoradiation Before Placebo (N=117) | Tarceva (N=77) | Placebo (N=75)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Allergic reaction/hypersensitivity (including drug fever)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Supraventricular and nodal arrhythmia Atrial fibrillation
Cardiac General - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constitutional symptoms - Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Skin - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Chest/Thorax (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Abdomen NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — None otherwise specified (NOS)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Thrombosis/ thrombus/ embolism

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No